CLINICAL TRIAL: NCT06637215
Title: Open, Parallel, Randomized Controlled, Non-inferior, Phase III Clinical Research on the Treatment Model of Ambulatory Surgery for Colorectal Cancer
Brief Title: Clinical Research on the Treatment Model of Ambulatory Surgery for Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Kai Li, Deputy Director of surgical Oncology, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstHCMU_ambulatory_surgery
Record Dates: First submitted 2024-09-09; First posted 2024-10-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Carcinoma; Day Surgery
Keywords: Colorectal cancer; Day surgery; Laparoscope
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laparoscopic colorectal day surgery (Experimental): laparoscopic colorectal day surgery in patients with colorectal tumor who are generally in good health and have sufficient organ functions
  Interventions: Procedure: laparoscopic colorectal day surgery
- traditional laparoscopic colorectal surgery (Active Comparator): traditional laparoscopic colorectal surgery in patients with colorectal tumor who are generally in good health and have sufficient organ functions
  Interventions: Procedure: traditional laparoscopic colorectal surgery

INTERVENTIONS:
Procedure: laparoscopic colorectal day surgery — laparoscopic colorectal day surgery in patients with colorectal tumor who are generally in good health and have sufficient organ functions
  Arms: laparoscopic colorectal day surgery
Procedure: traditional laparoscopic colorectal surgery — traditional laparoscopic colorectal surgery in patients with colorectal tumor who are generally in good health and have sufficient organ functions
  Arms: traditional laparoscopic colorectal surgery

SUMMARY:
To investigate the postoperative complication incidence and long-term efficacy between ambulatory surgery for colorectal cancer and traditional laparoscopic colorectal surgery in patients with colorectal tumor who are generally in good health and have sufficient organ functions。

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined this study and signed an informed consent form；
2. Age: 18-75 years old；
3. The patient should have a good general condition and no serious internal medicine comorbidities (ASA classification of the American Anesthesiology Association is Grade I~III)；
4. Complete colonoscopy and colonoscopy biopsy, and the pathology is confirmed to be adenocarcinoma/high-level intraepithelial neoplasia；
5. Enhanced CT or MRI examination before surgery, indicating that the tumor diameter is ≤5.0 cm；
6. Preoperative staging: cT1-3NanyM0;
7. Strictly follow the colorectal day surgery plan, and micro-laparoscopic radical colorectal cancer treatment can be adopted；
8. There are no contraindications for abdominal wall nerve block anesthesia or non-opiate analgesic drugs;
9. Does not require conventional anticoagulant therapy or antiplatelet therapy；
10. Relatives or co-residents should be able to provide 24 hours of full escort within at least 72 hours after the operation, the place of residence is not more than a 30-minute drive from the hospital, and they can understand and follow the phased treatment plan of diet, analgesic drugs, etc. after the operation.

Exclusion Criteria:

1. Elderly patients with multiple basic diseases；
2. Moderate to severe anemia；
3. Severe hypoproteinemia；
4. Diabetes that is not well controlled；
5. Contraindications to laparoscopic surgery；
6. Cases of emergency surgery due to acute intestinal obstruction, perforation or bleeding；
7. Patients with distant metastases；
8. Patients who are unwilling to sign informed consent or follow-up according to the research plan；
9. People with a history of psychotropic drug abuse and unable to quit or have mental disorders；
10. Patients who live alone or in psychosocial isolation, patients who cannot understand the postoperative nursing process；
11. After the operation, the place of residence is far away from the treated hospital or patients with insufficient medical resources and inconvenient transportation；
12. According to the judgment of the researcher, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the patient's research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (DFS) | From enrollment to the end of treatment at 36 months
Overall survival (OS) | From enrollment to the end of treatment at 36 months

SECONDARY OUTCOMES:
BIood system disorders | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  Anemia:
  Grade 1: HemogIobin (Hgb) <LLN - 10.0 g/dL; <LLN - 6.2 mmoI/L; <LLN - 100 g/L; Grade 2: Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmoI/L; <100 - 80g/L; Grade 3: Hgb <8.0 - 6.5 g/dL; <4.9 - 4.0 mmoI/L; <80 - 65g/L; transfusion indicated; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death.
Pain evaluation | From one hour after surgery to the end of treatment at 48 hours
  Visual analogue scale (VAS) Using a ruler with 10 scales, and the two ends of the ruler are "0" and "10". 0 points indicate painless, and 10 points represent the most severe pain that is unbearable.
  The patients mark the corresponding position on the ruler that can represent the degree of pain. The doctor assigns a score to the patient based on the position marked by the patient. 2-4 points represent mild pain, 5-7 points represent moderate pain, and 8-9 points represent severe pain.
Cardiac disorders | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  Acute coronary syndrome Grade 1: - Grade 2: symptomatic, progressive angina; cardiac enzymes normaI; hemodynamicaIIy stabIe; Grade 3: symptomatic, unstabIe angina and/or acute myocardiaI infarction, cardiac enzymes abnormaI, hemodynamicaIIy stabIe; Grade 4: symptomatic, unstabIe angina and/or acute myocardiaI infarction, cardiac enzymes abnormaI, hemodynamicaIIy unstabIe.
  Grade 5: Death.
CoIonic fistuIa | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  Grade 1: Asymptomatic; cIinicaI or diagnostic observations onIy; intervention not indicated; Grade 2: symptomatic; aItered gastrointestinaI function; Grade 3: severeIy aItered GI function; boweI rest, TPN or hospitaIization indicated; eIective operative intervention indicated; Grade 4: Life-threatening; Grade 5: Death.
AbdominaI infection | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  AbdominaI infection Grade 1: - Grade 2: - Grade 3: IV antibiotic, antifungaI, or antiviraI intervention indicated; radioIogic or operative intervention indicated; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death.
AnorectaI infection | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  AnorectaI infection Grade 1: LocaIized; IocaI intervention indicated; Grade 2: OraI intervention indicated (e.g. , antibiotic, antifungaI, antiviraI); Grade 3: IV antibiotic, antifungaI, or antiviraI intervention indicated; radioIogic, endoscopic, or operative intervention indicated; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death.
Fever | From enrollment to the end of treatment at 1 week
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe but not immediately life-threatening; Grade 4: Life-threatening; Grade 5: Death.
  Fever Grade 1: 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F); Grade 2: >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F); Grade 3: >40.0 degrees C (>104.0 degrees F) for <=24 hrs; Grade 4: >40.0 degrees C (>104.0 degrees F) for >24 hrs; Grade 5: Death.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No